CLINICAL TRIAL: NCT01379625
Title: Phase 2 Study of Triheptanoin for Treatment of Long-Chain Fatty Acid Oxidation Disorders
Brief Title: Study of Triheptanoin for Treatment of Long-Chain Fatty Acid Oxidation Disorder
Acronym: Triheptanoin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Melanie B Gillingham, Assistant Professor, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FD003895
Record Dates: First submitted 2011-06-21; First posted 2011-06-23 (Estimated); Results first posted 2017-03-23 (Actual); Last update posted 2017-03-23 (Actual); Status verified 2017-03

CONDITIONS: Very Long-chain acylCoA Dehydrogenase (VLCAD) Deficiency; Carnitine Palmitoyltransferase 2 (CPT2) Deficiency; Mitochondrial Trifunctional Protein (TFP) Deficiency; Long-chain 3 hydroxyacylCoA Dehydrogenase (LCHAD) Deficiency
Keywords: fatty acid oxidation; triheptanoin; long-chain fatty acid oxidation disorders; LCHADD; VLCADD; CPT2; TFP
MeSH Terms: conditions — VLCAD deficiency | interventions — triheptanoin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Medium Chain Triglyceride (MCT) (Active Comparator): Subjects randomized to consume 20% of energy from MCT
  Interventions: Drug: Triheptanoin
- Triheptanoin (Experimental): Subject randomized to consume 20% of energy from triheptanoin.
  Interventions: Drug: Triheptanoin

INTERVENTIONS:
Drug: Triheptanoin — Triglyceride with three heptanoin or 7 carbon fatty acids esterified to a glycerol backbone
  Other Names: IND 113386; C7

SUMMARY:
Humans eat long-chain fat in their diet and use it for energy during exercise and during periods of fasting. Patients with long-chain fatty acid oxidation disorders cannot use dietary fat for energy. They sometimes develop muscle breakdown, and severe pain with exercise or illness. They can also develop a heart that does not function properly. These patients are tired and expend less energy than people who do not have a long-chain fatty acid oxidation disorder. However, they can use a supplement oil called medium chain triglyceride or MCT. This study will determine if a new experimental oil called Triheptanoin can decrease the muscle pain and increase the heart function and the amount of energy in patients with long-chain fatty acid oxidation disorders. Funding source - FDA's OOPD

DETAILED DESCRIPTION:
Recruitment: Patients with a long-chain fatty acid oxidation disorder will be recruited through our clinic, past research participants, a patient support website, and recruitment letters mailed to physicians around the US. We will enroll 16 subjects at OHSU and 16 subjects at the University of Pittsburgh, age 7 to 40, with a disorder in fatty acid oxidation.

Procedures: Subjects will be admitted to the clinical research center for 4 days. They will collect all their urine for 24 hours. Heart function will be measured using ultrasound an electrocardiogram (ECG). The motion of the heart will be measured by magnetic resonance imaging (MRI). For this test, the patient lies in the magnetic field of the MRI machine in the Advanced Imaging Resource Center (AIRC) for about 45 minutes. The amount of muscle and fat in the whole body and inside the liver and muscle will be measured by MRS and by dual X-ray absorptiometry (DEXA). Subjects will walk on a treadmill for about 45 minutes. The amount of Calories they use, their heart rate, and if they burn fat or carbohydrates will be measured. Blood samples will be collected before and after exercise. A meal test will be used to determine how much fat they burn. The subjects will drink a liquid breakfast with a stable isotope labeled fat in the breakfast. Breath and blood samples will be collected before and after the meal. The amount Calories burned by each subject will be measured when they are at rest on a bed by indirect calorimetry. The amount of Calories burned by subjects when they are doing their routine daily activities will be measured at home by doubly labeled water. All of these tests will be done at baseline. Then, subjects will be randomly assigned to consume MCT (current standard of care) or triheptanoin at 20% of their estimated Calorie needs for 4 months. The subject and/or the parent will be taught how to use the supplement oil in their diet for cooking and baking. The subject will be sent home and the oil will be shipped to their home. The study coordinator will call the subject or subject's guardian each week to monitor the subject's diet, potential side effects and assist with diet planning. At the end of 4 months, all of the baseline tests will be repeated.

Triheptanoin is experimental oil. It is a clear, odorless oil that can be mixed with foods and used in cooking. Almost all oils are made from even chains of carbon molecules. Triheptanoin is different because the carbon chains are odd in number. The co-investigator of this study at the University of Pittsburgh, Dr. Jerry Vockely, holds an IND for the prescription, and use of triheptanoin in humans (IND 106011).

Data Analysis: The change in exercise ability, heart function, Calories used and body fat after 4 months will be compared between subjects randomized to MCT versus triheptanoin.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of Very long-chain acylCoA dehydrogenase (VLCAD) Deficiency, Carnitine Palmitoyltransferase 2 (CPT2) Deficiency, Mitochondrial Trifunctional Protein (TFP) Deficiency, or Long-chain 3 hydroxyacylCoA dehydrogenase (LCHAD) deficiency
* > 7 years
* Ability to travel to CRC to participate
* Ability to follow protocol

Exclusion Criteria:

* Hgb < 10 g/dl
* Peripheral neuropathy that limits ability to complete treadmill studies
* Inclusion in another research study that alters macronutrient intake
* Pregnant females
* history of myocardial infarction or cardiovascular disease

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2011-09; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melanie B Gillingham, PhD, Principal Investigator — Oregon Health and Science University
Locations (2):
- United States (2):
  - Oregon Health & Science University, Portland, Oregon
  - University of Pittsburgh, Pittsburgh, Pennsylvania

REFERENCES:
- [Derived] Gillingham MB, Heitner SB, Martin J, Rose S, Goldstein A, El-Gharbawy AH, Deward S, Lasarev MR, Pollaro J, DeLany JP, Burchill LJ, Goodpaster B, Shoemaker J, Matern D, Harding CO, Vockley J. Triheptanoin versus trioctanoin for long-chain fatty acid oxidation disorders: a double blinded, randomized controlled trial. J Inherit Metab Dis. 2017 Nov;40(6):831-843. doi: 10.1007/s10545-017-0085-8. Epub 2017 Sep 4. PMID 28871440

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Medium Chain Triglyceride (MCT) | Triheptanoin
Started | 16 | 16
Completed | 16 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Subjects were 7 years of age or greater with one of 3 fatty acid oxidation disorders: CPT2, VLCAD or LCHAD/TFP.
Groups:
- Total: Total of all reporting groups
Arm/Group | Medium Chain Triglyceride (MCT) | Triheptanoin | Total
Number analyzed (Participants) | 16 | 16 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.3 (12.7) | 27.2 (15.9) | 24.8 (14.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 6 | 6 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 15 | 16 | 31
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 16 | 16 | 32
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 16 | 16 | 32
Body Weight [Mean (Standard Deviation); unit: kilograms] | 67.1 (26.8) | 62.1 (23.5) | 64.6 (24.9)
Ejection Fraction [Mean (Standard Deviation); unit: percent] — Echocardiogram ejection fraction as a %. This was not completed for all the participant. There were 11 participants in the MCT group and 10 participants in the Triheptanoin group who are included in this baseline measure. Population: There was a change in the protocol from cardiac MRI to echo after the 1st 7 participants and some of the echocardiogram results were unreadable due to technical errors. A total of 11 subjects in the MCT and 10 subjects in triheptanoin group were analyzed.
  percent
    number analyzed (Participants) | 11 | 10 | 21
    (all) | 63 (5.3) | 57 (9.2) | 59.7 (8.0)
Exercise Heart Rate [Mean (Standard Deviation); unit: beats per minute] — All participants performed a moderate intensity exercise treadmill walking at an estimated 60% of their estimated max heart rate for 40 minutes. The exercise heart rate at minute 30 when the exercise was steady is reported.
  beats per minute | 132 (7) | 125 (12) | 128 (10)
Total Energy Expenditure [Mean (Standard Deviation); unit: kcal/day] — Total energy expenditure in kcal/day was measured by doubly labled water in 12 subjects in the MCT group and in 13 of the subjects in the Triheptanoin group. Population: One participant in the MCT group and one participant in the Triheptanoin group did not return their urine samples for the doubly labeled water analysis. A total of 15 in each group were analyzed.
  kcal/day
    number analyzed (Participants) | 15 | 15 | 30
    (all) | 2567 (604) | 2230 (512) | 2392 (572)

OUTCOME MEASURES:

1. Primary Outcome: Energy Expenditure
Description: Total energy expenditure will be measured by doubly labeled water and resting energy expenditure will be measured by indirect calorimetry at baseline and again after 4 months of either MCT or trihpetanoin treatment.
Time Frame: change from baseline after 4 months of treatment
Population: One subject in each group did not complete the doubly labeled water measures. A total of 15 in each group measured total energy expenditure at baseline and at the end of the study. This value compares the change over treatment.
Measure: Mean (Standard Deviation); unit: kcal/day
Arm/Group | Medium Chain Triglyceride (MCT) | Triheptanoin
Number analyzed (Participants) | 15 | 15
kcal/day | -73 (335) | 107 (387)

2. Primary Outcome: Ejection Fraction
Description: Change in resting ejection fraction over 4 month treatment period
Time Frame: 4 months
Population: Change in resting ejection fraction over 4 month treatment period calculated as: 4 month ejection fraction-baseline ejection fraction. Only participants with available data are included in this analysis.
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Medium Chain Triglyceride (MCT) | Triheptanoin
Number analyzed (Participants) | 11 | 10
percent | -1.91 (4.16) | 2.14 (4.43)

3. Secondary Outcome: Exercise Heart Rate
Description: Subjects will complete a submaximal treadmill exercise study at baseline. Exercise heart heart, ventilation and perceived exertion will be measured. Subjects will be randomized to MCT or triheptanoin supplementation for 4 months. At the end of treatment, the exercise test will be repeated keeping work performed constant. Change in exercise heart rate, ventilation and exertion will be compared between groups.
Time Frame: change from baseline to 4 months of treatment
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Medium Chain Triglyceride (MCT) | Triheptanoin
Number analyzed (Participants) | 16 | 16
beats per minute | -0.1 (9.6) | -12.6 (34)

ADVERSE EVENTS:
Time Frame: Four months
Arm/Group | Medium Chain Triglyceride (MCT) | Triheptanoin
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 12/16 | 11/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Medium Chain Triglyceride (MCT) (N=16) | Triheptanoin (N=16)
Gastrointestinal Upset (Gastrointestinal disorders) | 12 (38) | 11 (24) — Gastrointestinal Upset including stomach pain, burning, or cramping.
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 4 (7) | 5 (7) — Acute rhabdomyolysis requiring hospitalization is expected. This is a known complication of fatty acid oxidation disorders.
Diarrhea/Loose stools (Gastrointestinal disorders) | 6 (12) | 5 (9) — Report of diarrhea or loose stools during the treatment period.
muscle pain/ elevated CPK (Musculoskeletal and connective tissue disorders) | 10 (18) | 11 (16) — This is an anticipated adverse event because muscle pain with elevated CPK is a complication of a fatty acid oxidation disorder.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No